CLINICAL TRIAL: NCT03907722
Title: The 3q25 rs2305619 Polymorphism is Associated With Coronary Microvascular Obstruction Following Primary Angioplasty for Acute ST-segment Elevation Myocardial Infarction
Brief Title: The 3q25 rs2305619 Polymorphism Associates With Microvascular Obstruction in STEMI
Status: Completed | Type: Observational
Sponsor: Indonesian Cardiovascular Research Center (Other)
Responsible Party: Principal Investigator, Surya Dharma, Principal Investigator, Indonesian Cardiovascular Research Center
Other Study IDs: IndonesianCRC2
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: STEMI; Microvascular Coronary Artery Disease
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — PTX3 protein

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genotypic variants: AA, AG and GG genotype
  Interventions: Other: Long pentraxin 3

INTERVENTIONS:
Other: Long pentraxin 3 — Primary PCI

SUMMARY:
The investigators enrolled 217 patients with acute STEMI undergoing primary PCI. The rs2305619 polymorphism was evaluated by real time PCR and plasma PTX3 concentration was assessed by human PTX3 ELISA kit.

DETAILED DESCRIPTION:
The investigators enrolled 217 patients with acute STEMI undergoing primary PCI in a tertiary care academic cardiovascular center. The rs2305619 polymorphism was evaluated by real time PCR and plasma PTX3 concentration was assessed by human PTX3 ELISA kit. The primary outcome of the study was the incidence of coronary microvascular obstruction defined as thrombolysis in myocardial infarction (TIMI) grade <3 flow after primary PCI or TIMI grade 3 flow with myocardial blush grade 0 or 1. Patients were grouped based on the genotypic variants (AA, AG and GG). The primary outcome was compared among the three variants, as well as the PTX3 concentration and 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute STEMI with symptom onset <12 h and treated by primary PCI

Exclusion Criteria:

* STEMI patients who received fibrinolytic therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with STEMI symptom onset <12h admitted to the ED and planned for primary PCI
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Incidence of microvascular obstruction | Immediate after pci
  Percentage

SECONDARY OUTCOMES:
Incidence of mortality | 30 days
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Surya Dharma, MD, PhD, Principal Investigator — Indonesian Cardiovascular Center
Locations (1):
- Indonesian Cardiovascular Research Center, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No